CLINICAL TRIAL: NCT02246374
Title: A Randomized Feasibility Clinical Trial of the Management of the Medically-Refractory Motor Symptoms of Advanced Idiopathic Parkinson's Disease With Unilateral Lesioning of the Subthalamic Nucleus Using the ExAblate Transcranial System
Brief Title: ExAblate Transcranial MRgFUS of the Subthalamic Nucleus for Treatment of Parkinson's Disease
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: PD003
Record Dates: First submitted 2014-09-18; First posted 2014-09-22 (Estimated); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease; ExAblate; MRgFUS
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ExAblate Treated Arm (Experimental): ExAblate Transcranial System subthalamotomy for motor symptoms of Parkinson's Disease.
  Interventions: Device: ExAblate Transcranial System
- ExAblate Sham Treated Arm (Sham Comparator): ExAblate Transcranial System sham subthalamotomy for motor symptoms of Parkinson's Disease. Sham subjects completing the 4 Month visit may be offered the actual ExAblate subthalamotomy.
  Interventions: Device: ExAblate Transcranial System

INTERVENTIONS:
Device: ExAblate Transcranial System — ExAblate Transcranial System subthalamotomy for symptoms of Parkinson's Disease
  Other Names: MRgFUS; FUS; Focused Ultrasound; MR Guided Focused Ultrasound

SUMMARY:
This is primarily a safety protocol to evaluate the safety of subthalamotomy using Transcranial ExAblate for treatment of Parkinson's Disease (PD) motor features.

DETAILED DESCRIPTION:
This study is designed as a prospective, randomized, double-blind (to subjects and examiners), two-arm (ExAblate treated arm vs ExAblate Sham treated control arm) feasibility study. All treated subjects will be followed for 12 months.

Data will be collected to establish the basic safety and clinical efficacy of this type of treatment as the basis for later studies that will evaluate the full clinical efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women, age 30 years and older
2. Subjects who are able and willing to give informed consent and able to attend all study visits
3. Subjects with a diagnosis of idiopathic PD by UK Brain Bank Criteria as confirmed by a movement disorder neurologist at the site
4. Levodopa responsive as defined by at least a 30% reduction in MDS-UPDRS motor sub-scale in the ON vs OFF medication state
5. Disabling motor clinical features not optimally controlled by an adequate medication prescription. An adequate medication prescription is defined as a therapeutic dose of each medication or the development of side effects as the medication dose is titrated
6. Predominant disability from one side of the body (i.e unilateral or markedly asymmetric disease) as determined by movement disorders neurologist and neurosurgeon
7. Subjects should be on a stable dose of all PD medications for 30 days prior to study entry
8. Subthalamic nucleus is visible on MRI so that it can be targeted by the ExAblate device
9. Subjects should have a Screening motor assessment of ≥ 35 while OFF medications on the MDS-UPDRS
10. Subject is able to communicate sensations during the ExAblate Transcranial procedure

Exclusion Criteria:

1. Hoehn and Yahr stage in the ON medication state of 2.5 or greater
2. Presence of severe dyskinesia as noted by a score of 3 or 4 on questions 4.1 and 4.2 of the MDS-UPDRS
3. Presence of other central neurodegenerative disease suspected on neurological examination. These include: multisystem atrophy, progressive supranuclear palsy, corticobasal syndrome, dementia with Lewy bodies, and Alzheimer's disease
4. Any suspicion that Parkinsonian symptoms are a side effect from neuroleptic medications
5. Subjects who have had deep brain stimulation or a prior stereotactic ablation of the basal ganglia
6. Presence of significant cognitive impairment defined as score ≤ 21 on the Montreal Cognitive Assessment (MoCA) or Mattis Dementia Rating Scale of 120 or lower
7. Unstable psychiatric disease, defined as active uncontrolled depressive symptoms, psychosis, delusions, hallucinations, or suicidal ideation. Subjects with stable, chronic anxiety or depressive disorders may be included provided their medications have been stable for at least 60 days prior to study entry and if deemed appropriately managed by the site neuropsychologist
8. Subjects with significant depression as determined following a comprehensive assessment by a neuropsychologist. Significant depression is being defined quantitatively as a score of greater than 14 on the Beck Depression Inventory
9. Legal incapacity or limited legal capacity as determined by the neuropsychologist
10. Subjects exhibiting any behavior(s) consistent with ethanol or substance abuse as defined by the criteria outlined in the DSM-IV as manifested by one (or more) of the following occurring within the preceding 12 month period:

    1. Recurrent substance use resulting in a failure to fulfill major role obligations at work, school, or home (such as repeated absences or poor work performance related to substance use; substance-related absences, suspensions, or expulsions from school; or neglect of children or household)
    2. Recurrent substance use in situations in which it is physically hazardous (such as driving an automobile or operating a machine when impaired by substance use)
    3. Recurrent substance-related legal problems (such as arrests for substance related disorderly conduct)
    4. Continued substance use despite having persistent or recurrent social or interpersonal problems caused or exacerbated by the effects of the substance (for example, arguments with spouse about consequences of intoxication and physical fights)
11. Subjects with unstable cardiac status including:

    1. Unstable angina pectoris on medication
    2. Subjects with documented myocardial infarction within six months of protocol entry
    3. Significant congestive heart failure defined with ejection fraction < 40
    4. Subjects with unstable ventricular arrhythmias
    5. Subjects with atrial arrhythmias that are not rate-controlled
12. Severe hypertension (diastolic BP > 100 on medication)
13. History of or current medical condition resulting in abnormal bleeding and/or coagulopathy
14. Receiving anticoagulant (e.g. warfarin) or antiplatelet (e.g. aspirin) therapy within one week of focused ultrasound procedure or drugs known to increase risk or hemorrhage (e.g. Avastin) within one month of focused ultrasound procedure
15. Subjects with risk factors for intraoperative or postoperative bleeding as indicated by: platelet count less than 100,000 per cubic millimeter, a documented clinical coagulopathy, or INR coagulation studies exceeding the institution's laboratory standard
16. Patient with severely impaired renal function with estimated glomerular filtration rate <30 mL/min/1.73m2 (or per local standards should that be more restrictive) and/or who is on dialysis
17. Subjects with standard contraindications for MR imaging such as non-MRI compatible implanted metallic devices including cardiac pacemakers, size limitations, etc.
18. Significant claustrophobia that cannot be managed with mild medication
19. Subjects who weigh more than the upper weight limit of the MR table and who cannot fit into the MR scanner
20. Subjects who are not able or willing to tolerate the required prolonged stationary supine position during treatment
21. History of intracranial hemorrhage
22. History of multiple strokes, or a stroke within past 6 months
23. Subjects with a history of seizures within the past year
24. Subjects with brain tumors
25. Subjects with intracranial aneurysms requiring treatment or arterial venous malformations (AVMs) requiring treatment
26. Are participating or have participated in another clinical trial in the last 30 days
27. Any illness that in the investigator's opinion preclude participation in this study
28. Subjects unable to communicate with the investigator and staff
29. Pregnancy or lactation
30. Subjects who have an overall Skull Density Ration lower than 0.40 as calculated from the screening CT

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2014-09; Primary Completion 2026-06 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence and severity of adverse events | Baseline to 4 months post treatment
  Safety will evaluate the incidence and severity of adverse events associated with ExAblate subthalamotomy for the treatment of Parkinson's Disease motor features.
Mean change in MDS-UPDRS Part III scores | Baseline to 4 months post treatment
  This is a feasibility trial with no hypothesis testing. Primary efficacy will be evaluated using basic summary statistics including comparison of between- and within-group differences in the mean change (from baseline to 4 months) of the motor MDS-UPDRS Part III score for the side contralateral to subthalamotomy in the off-medication condition.

SECONDARY OUTCOMES:
Long Term Adverse Events Profile | Baseline to 12- months post treatment
  Additional safety will be evaluated by follow up of adverse events through 12 months post treatment.

OTHER OUTCOMES:
Mean change in MDS-UPDRS total score | Baseline to 12- months post treatment
  Duration of outcomes will be further evaluated using the MDS-UPDRS total score
Mean change in MDS-UPDRS Part IV scores | Baseline to 12-months post treatment
  Long term impact of ExAblate transcranial pallidotomy will be further evaluated using the MPS-UPDRS Part IV scores

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Elias, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States